CLINICAL TRIAL: NCT06133010
Title: A Phase 2, Observer-Blind, Placebo-Controlled, Proof-of-Concept Trial to Evaluate the Efficacy, Safety, and Immunogenicity of mRNA-1647 Cytomegalovirus Vaccine in Liver Transplant Candidates and Recipients
Brief Title: A Study of mRNA-1647 Cytomegalovirus Vaccine in Liver Transplant Candidates and Recipients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was cancelled by Sponsor
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1647-P206
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cytomegalovirus Infection
Keywords: mRNA-1647; Vaccine; Liver Transplant; CMV; Human Herpesvirus; Cytomegalovirus Vaccine; Cytomegalovirus Infections; Cytomegalovirus Disease; Cytomegalovirus; Virus Disease; Infection Viral; DNA Virus Infections; Messenger RNA
MeSH Terms: conditions — Cytomegalovirus Infections; Herpes Simplex; Virus Diseases; DNA Virus Infections | interventions — mRNA-1647 cytomegalovirus vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1647 (Experimental): CMV-seronegative and CMV-seropositive participants will receive 3 intramuscular (IM) injections of mRNA-1647 vaccine on Days 1, 29, and 57.
  Interventions: Biological: mRNA-1647
- Placebo (Experimental): CMV-seronegative and CMV-seropositive participants will receive 3 IM injections of mRNA-1647 vaccine-matching placebo on Days 1, 29, and 57.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1647 — Sterile liquid for injection
  Arms: mRNA-1647
Biological: Placebo — Sterile liquid for injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of pre-transplant mRNA-1647 on post-transplant cytomegalovirus (CMV) virologic outcomes, anti-CMV antiviral use, and clinical outcomes in CMV-seropositive and CMV-seronegative liver transplant candidates who receive transplants and to assess the safety, reactogenicity, and immunogenicity of mRNA-1647 in all participants.

ELIGIBILITY:
Inclusion Criteria:

* Having a negative (that is, CMV-seronegative) or a positive (that is, CMV-seropositive) result using a blood IgG assay performed at the central laboratory or a previously documented seropositive result.
* Listed and anticipated to receive their first deceased donor or living donor liver transplant within 2 months to 12 months of enrollment.
* A person of nonchildbearing potential, as defined in the protocol.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection, and agreement to continue adequate contraception or abstinence through 3 months following last study injection.

Exclusion Criteria:

* Listed as "status 1A" for liver transplant.
* Hypersensitivity to acyclovir, ganciclovir, or valganciclovir.
* Previous receipt of a solid organ or hematopoietic transplant.
* Listed for or anticipated to receive an organ transplant other than liver, either simultaneously or sequentially.
* Receipt of prior investigational CMV vaccines or participation in another CMV therapeutic study that may interfere with study outcome measures as determined by the Investigator.
* Suspected or known allergic reaction to any component of any mRNA vaccine, including mRNA-1647, or its excipients.
* Human immunodeficiency virus (HIV) infection (based on documented testing performed during the transplant evaluation process and no clinical suspicion of HIV infection).
* Prior (ever) receipt of a stem cell transplant (peripheral blood stem cell, marrow, cord blood).
* Any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2027-02-14 (Estimated); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
Post-transplant: Time to the First Occurrence of a Clinically Significant Cytomegalovirus Infection (CS-CMVi) In Seropositive Participants | Day 373 through Day 466
  CS-CMVi will be defined as CMV viremia necessitating treatment (with treatment initiated at viral load ≥250 international units/milliliter [IU/mL] and/or CMV disease) through Day 466.
Number of Participants With Solicited Local and Systemic Adverse Reactions | Up to Day 64 (7 days after the last study injection)
Number of Participants With Unsolicited Adverse Events | Up to Day 87 (28 days after the last study injection)
Number of Participants With Medically Attended Adverse Events | Up to Day 237 (6 months after the last study injection)
Number of Participants With Serious Adverse Events | Day 1 through Day 542
Number of Participants With Adverse Events of Special Interest | Day 1 through Day 542
Number of Participants With Adverse Events Leading to Discontinuation | Day 1 through Day 542

SECONDARY OUTCOMES:
Post-transplant: Time to First Occurrence of Adjudicated CMV Disease in Seronegative Participants Who Receive a Liver Transplant from a CMV-seropositive Donor | Day 373 through Day 466
  Evidence of adjudicated CMV disease and/or infection, as defined in the protocol, will include signs, symptoms, and biopsy evidence.
Post-transplant: Number of Seronegative Participants Who Received a Liver Transplant from a CMV-seropositive Donor with Any Occurrence of CMV Viremia | Day 373 through Day 466
  Viremia will be defined as any detectable viral load through Day 466.
Post-transplant: Number of Seronegative Participants Who Received a Liver Transplant from a CMV-seropositive Donor with an Occurrence of CMV Viremia | Day 373 through Day 466
  Viremia will be defined as a viral load ≥1000 IU/mL through Day 466.
Post-transplant: Duration of anti-CMV Antiviral Therapy | Day 373 through Day 466
Post-transplant: Time to Initiation of anti-CMV Antiviral Therapy | Day 373 through Day 466
Post-transplant: Number of Participants Requiring anti-CMV Antiviral Therapy | Day 373 through Day 466
Number of Participants With Investigator-reported CMV Disease | Day 380 through Day 466
  Evidence of CMV disease and/or infection, as defined in the protocol, will include signs, symptoms, and biopsy evidence.
Number of Seropositive Participants With CMV Disease, Defined as Adjudicated CMV Disease | Day 380 through Day 466
  Evidence of adjudicated CMV disease and/or infection, as defined in the protocol, will include signs, symptoms, and biopsy evidence. Adjudication will occur by a blinded adjudication committee per protocol.
Post-transplant: Time to Onset of Initial CMV Viremia | Day 373 through Day 466
Post-transplant: Duration of Initial CMV Viremia | Day 373 through Day 466
Post-transplant: Number of Participants With Recurrent CMV Viremia Following 2 Consecutive Undetectable CMV Viral Load Assays | Day 373 through Day 466
  Recurrent CMV viremia will be defined as a viral load ≥250 IU/mL for seropositive participants and any detectable level for seronegative participants who receive a seropositive organ.
Post-transplant: Duration of Recurrent CMV Viremia | Day 373 through Day 466
  Recurrent CMV viremia will be defined as a viral load ≥250 IU/mL for seropositive participants and any detectable level for seronegative participants who receive a seropositive organ
Post-transplant: Peak Viral Load in Participants with CMV Viremia | Day 373 through Day 466
Post-transplant: CMV Viremia Area Under the Curve | Day 373 through Day 466
Post-transplant: Number of Participants With Neutropenia | Day 373 through Day 466
  Neutropenia will be defined as an absolute neutrophil count ≤500 absolute neutrophils/microliter.
Post-transplant: Number of Participants With Leukopenia on 2 Successive Measurements Separated by at Least 24 Hours | Day 365 through Day 466
  Leukopenia will be defined as an absolute white blood cells (WBC) <3500 cells/cubic milliliter (mm^3) if baseline was ≥4000 cells/mm^3 or a decrease in WBC of >20% if the baseline count was <4000 cells/mm^3.
Post-transplant: Number of Participants Requiring Liver Re-transplantation | Day 365 through Day 542
Post-transplant: All-cause Mortality | Day 365 through Day 542
Post-transplant: Number of Participants with Biopsy Proven Allograft Rejection | Day 365 through Day 542
  Biopsy proven allograft rejection will be adjudicated by a blinded adjudication committee per protocol.
Pre-transplant: Titer of CMV- Specific Neutralizing Antibody (nAb) as Measured by Cell-based Neutralization Assay | Day 1, Day 29, Day 57, Day 87, Day 237, and Day 365
Post-transplant: Titer of CMV-Specific nAb Post-transplant as Measured by Cell-based Neutralization Assay | Day 365, Day 466, and Day 542
Pre- and Post-transplant: Geometric Mean Titer (GMT) of Anti-glycoprotein B (gB)-specific Immunoglobulin G (IgG) and Antipentamer-specific IgG as Measured by Enzyme-linked Immunosorbent Assay (ELISA) | Day 1, Day 29, Day 57, Day 87, Day 237, Day 365, Day 466, and Day 542
Pre- and Post-transplant: Geometric Mean Concentration (GMC) of Anti-gB-specific IgG and Antipentamer-specific IgG as Measured by ELISA | Day 1, Day 29, Day 57, Day 87, Day 237, Day 365, Day 466, and Day 542
Pre- and Post-transplant: Geometric Mean Ratio (GMR) of Post-baseline/Baseline GMTs and GMCs | Day 1, Day 29, Day 57, Day 87, Day 237, Day 365, Day 466, and Day 542
Pre- and Post-transplant: Geometric Mean Fold Rise (GMFR) of Post-baseline/Baseline GMTs or GMCs | Day 1, Day 29, Day 57, Day 87, Day 237, Day 365, Day 466, and Day 542